CLINICAL TRIAL: NCT05589805
Title: Comparison of the Effectiveness of Low-intensity Laser and ESWT Treatments in Carpal Tunnel Syndrome
Brief Title: Comparison of Low-intensity Laser and ESWT in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif yaksi, Medical Doctor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-EY-07
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; extracorporeal shock wave therapy; laser treatment
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy; Laser Therapy; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT group (Experimental): In addition to wrist splint, ESWT treatment (1.5 bar, 5Hz, 1000 beats) will be applied to the patients with the Elmed Vibrolith Ortho brand ESWT device, which we routinely use in the treatment of carpal tunnel syndrome, for 3 weeks, once a week.
  Interventions: Device: Extracorporeal shock wave therapy
- Laser group (Experimental): In addition to the wrist splint, the patients will be treated with the BTL-4110 Laser Topline model low-intensity laser device, which we routinely use in the treatment of carpal tunnel syndrome in our hospital, 5 days a week for 15 sessions of laser treatment.
  Interventions: Device: Laser therapy
- Control group (Active Comparator): Patients will only be given a wrist splint to keep the wrist in neutral position.
  Interventions: Other: Control group

INTERVENTIONS:
Device: Extracorporeal shock wave therapy — In addition to wrist splint, ESWT treatment (1.5 bar, 5Hz, 1000 beats) will be applied to the patients with Elmed Vibrolith Ortho brand ESWT device, which we routinely use in the treatment of carpal tunnel syndrome, for 3 weeks, once a week.
  Arms: ESWT group
Device: Laser therapy — In addition to the wrist splint, the patients will be treated with the BTL-4110 Laser Topline model low-intensity laser device, which we routinely use in the treatment of carpal tunnel syndrome in our hospital, 5 days a week for 15 sessions of laser treatment.
  Arms: Laser group
Other: Control group — Patients will only be given a wrist splint to keep the wrist in neutral position.
  Arms: Control group

SUMMARY:
Carpal tunnel syndrome is the most common neuropathy of the median nerve. Conservative methods are used in mild and moderate CTS in the treatment. In this study, we aimed to compare the effectiveness of low-intensity laser and ESWT treatments in patients with mild and moderate carpal tunnel syndrome diagnosed with EMG.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is the most common neuropathy of the median nerve. Its incidence increases between the ages of 40-60. Its prevalence is 4-5%, and incidence is 2.7%. It is more common in women than men. The vast majority of cases are idiopathic.The first symptoms usually start at night. The patient wakes up with a feeling of swelling without any visible swelling and symptoms such as burning, numbness and tingling in the median nerve region.In severe cases, hand weakness and thenar atrophy develop. Provocative tests such as phalen, reverse phalen, tinel, carpal compression test, tourniquet test can be used in the examination.The diagnosis of carpal tunnel syndrome is made by nerve conduction studies and electromyography. Conservative methods are used in mild and moderate CTS in the treatment. Surgical methods are recommended in severe cases and in cases unresponsive to conservative treatment.One of the methods used in the treatment is Laser (Light Amplification by Stimulated Emission of Radiation).There are low and high intensity laser applications according to their energy densities. The basic mechanism of action is tissue stimulation. ESWT (Extracorporeal Shock Wave Therapy), another treatment method, shows therapeutic properties by focusing high-amplitude sound waves on the desired area of the body. Apart from the mechanical effect, it also has an effect at the cellular level.In previous studies, both low-intensity laser and ESWT application were found to be effective in the treatment of carpal tunnel syndrome. However, as far as we know, there is no study comparing the efficacy of low-intensity laser therapy and ESWT therapy in carpal tunnel syndrome. In this study, we aimed to compare the effectiveness of low-intensity laser and ESWT treatments in patients with mild and moderate carpal tunnel syndrome diagnosed with EMG.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Having a clinic compatible with carpal tunnel syndrome,
* Patients with electrophysiological data compatible with mild and moderate carpal tunnel syndrome

Exclusion Criteria:

* Cervical radiculopathy , polyneuropathy , brachial plexopathy , thoracic outlet syndrome
* Regular use of oral steroids or nsaii in the last 3 months
* Systemic disease (DM, hypothyroidism, RA, gout, acromegaly, CKD, dialysis)
* Severe carpal tunnel syndrome (kts)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2023-10-20 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline
  It is a 10 cm line on the horizontal plane where the patient evaluates the pain. There are lines from 0 to 10. 0 means no pain, and 10 means very severe pain. After this information is given to the patient, the patient will mark the pain they feel within 1 week.
Visual Analog Scale | Post-treatment (3th week)
  It is a 10 cm line on the horizontal plane where the patient evaluates the pain. There are lines from 0 to 10. 0 means no pain, and 10 means very severe pain. After this information is given to the patient, the patient will mark the pain they feel within 1 week.
Boston Scale | Baseline
  The Boston Questionnaire was developed by Levine et al. in 1993. It consists of two parts, the symptom severity scale and the functional capacity scale.Boston Symptom Severity Scale consists of 11 questions. Symptoms such as pain, numbness, weakness, tingling are questioned. Symptoms are scored using a 5-answer scale between "absent and very severe". In the scoring of 11-55, a high score is interpreted as increased symptom severity.
  Boston Functional Capacity Scale consists of 8 questions. It questions the degree of difficulty of activities of daily living, and each question has five different answers with a score between 1 and 5. The average score is obtained by dividing the total score by the number of questions. Results are scored between 8-40 and high values are interpreted as impaired hand functionality.
Boston Scale | Post-treatment (3th week)
  The Boston Questionnaire was developed by Levine et al. in 1993. It consists of two parts, the symptom severity scale and the functional capacity scale.Boston Symptom Severity Scale consists of 11 questions. Symptoms such as pain, numbness, weakness, tingling are questioned. Symptoms are scored using a 5-answer scale between "absent and very severe". In the scoring of 11-55, a high score is interpreted as increased symptom severity.
  Boston Functional Capacity Scale consists of 8 questions. It questions the degree of difficulty of activities of daily living, and each question has five different answers with a score between 1 and 5. The average score is obtained by dividing the total score by the number of questions. Results are scored between 8-40 and high values are interpreted as impaired hand functionality.
Median nerve area measurement | Baseline
  It will be measured from the distal finger line by manually surrounding the nerve just below the hyperechoic line surrounding the median nerve with the ultrasound device.
Median nerve area measurement | Post-treatment (3th week)
  It will be measured from the distal finger line by manually surrounding the nerve just below the hyperechoic line surrounding the median nerve with the ultrasound device.
LANNS neuropathic pain scale | Baseline
  It is used to distinguish between neuropathic pain and nociceptive pain. It consists of 2 parts. The first part is filled by the patient. In the department, the physician tests whether allodynia is present. A score above 12 is classified as neuropathic pain.
LANNS neuropathic pain scale | Post-treatment (3th week)
  It is used to distinguish between neuropathic pain and nociceptive pain. It consists of 2 parts. The first part is filled by the patient. In the department, the physician tests whether allodynia is present. A score above 12 is classified as neuropathic pain.

SECONDARY OUTCOMES:
Visual Analog Scale (paresteshia) | Baseline
  t is a 10 cm line on the horizontal plane where the patient evaluates the pain. There are lines from 0 to 10. 0 means no pain, and 10 means very severe pain. After this information is given to the patient, the patient will mark the paresteshia they feel within 1 week.
Visual Analog Scale (paresteshia) | Post-treatment (3th week)
  t is a 10 cm line on the horizontal plane where the patient evaluates the pain. There are lines from 0 to 10. 0 means no pain, and 10 means very severe pain. After this information is given to the patient, the patient will mark the paresteshia they feel within 1 week.
Ouick Dash Score | Baseline
  There are 11 items in total in this questionnaire. It is evaluated between 1-5 points according to the increasing degree of symptoms or difficulty. At least 10 of the questions must be answered in order for the Quick DASH score to be calculated. The result of the calculation is evaluated between 0 and 100.0 is interpreted as no difficulty and no symptoms, 100 as no activity or severe symptoms.
Ouick Dash Score | Post-treatment (3th week)
  There are 11 items in total in this questionnaire. It is evaluated between 1-5 points according to the increasing degree of symptoms or difficulty. At least 10 of the questions must be answered in order for the Quick DASH score to be calculated. The result of the calculation is evaluated between 0 and 100.0 is interpreted as no difficulty and no symptoms, 100 as no activity or severe symptoms.

OTHER OUTCOMES:
Hand Grip Force | Baseline
  North Coast brand hydraulic hand dynamometer will be used. According to the standard position recommended by the American Association of Hand Therapists; Measurements are made when the patient is sitting upright, the knee angle is 90°, the shoulder is in adduction and neutral rotation, the elbow is in 90° flexion, the forearm is in midrotation, and the wrist is in neutral. 3 measurements are made, with a one-minute break between each measurement. The test result is taken as the average of the three measurements in kilograms.
Hand Grip Force | Post-treatment (3th week)
  North Coast brand hydraulic hand dynamometer will be used. According to the standard position recommended by the American Association of Hand Therapists; Measurements are made when the patient is sitting upright, the knee angle is 90°, the shoulder is in adduction and neutral rotation, the elbow is in 90° flexion, the forearm is in midrotation, and the wrist is in neutral. 3 measurements are made, with a one-minute break between each measurement. The test result is taken as the average of the three measurements in kilograms.
Finger Grip Force | baseline
  North Coast brand hydraulic pinchmeter will be used for finger grip strength measurement. It is evaluated in two different positions as atheral and pinch (triple) grip.
Finger Grip Force | Post-treatment (3th week)
  North Coast brand hydraulic pinchmeter will be used for finger grip strength measurement. It is evaluated in two different positions as atheral and pinch (triple) grip.